CLINICAL TRIAL: NCT01830582
Title: Pilot Study of Advanced MR Imaging for Early Biologic Tumor Changes to Neoadjuvant Chemoradiation Treatment for Rectal Cancer
Brief Title: Advanced MR Imaging for Early Biologic Tumor Changes to Neoadjuvant Chemoradiation Treatment for Rectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 13-019
Record Dates: First submitted 2013-04-10; First posted 2013-04-12 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Rectal Cancer
Keywords: MRI; rectum; 13-019
MeSH Terms: conditions — Rectal Neoplasms

ARMS (4):
- 1 A (Experimental): The patients will undergo the standard pre chemoradiation MRI scan, followed by a repeat research scan 24 hours (+/- 6 hours) after their first radiation treatment. Then they will get another research MRI scan during the second week (+/- 5 days) of radiation. Finally they will get a standard post chemoradiation MRI scan prior to surgery.
  Interventions: Procedure: Advanced MR Imaging
- 1 B (Experimental): The patient will undergo the standard pre chemoradiation MRI scan, followed by a repeat research scan 48 hours (+/- 6 hours) after their first radiation treatment. Then they will get another research MRI scan during the third week (+/- 5 days) of radiation. Finally they will get a standard post chemoradiation MRI scan prior to surgery.
  Interventions: Procedure: Advanced MR Imaging
- 1 C (Experimental): The patient will undergo the standard pre chemoradiation MRI scan, followed by a repeat research scan 72 hours (+/- 6 hours) after their first radiation treatment. Then they will get another research MRI scan during the fourth week (+/- 5 days) of radiation. Finally they will get a standard post chemoradiation MRI scan prior to surgery.
  Interventions: Procedure: Advanced MR Imaging
- 2 (Experimental): The last patient patients that will undergo a standard pre-chemoradiation MRI scan, followed by a repeat research scan either 24, 48 or 72 hours (+/- 6 hours) after their first radiation treatment. Then they will get another research MRI scan during the second, third or fourth week (+/- 5 days) of radiation. Finally they will get a standard post chemoradiation MRI scan prior to surgery.
  Interventions: Procedure: Advanced MR Imaging

INTERVENTIONS:
Procedure: Advanced MR Imaging

SUMMARY:
The purpose of this study is to see whether three new types of MRI techniques used during magnetic resonance imaging (MRI) of the pelvis to look at rectal cancer can help doctors to tell if the tumor is getting better in response to the radiation and/or chemotherapy treatments.

DETAILED DESCRIPTION:
This is a pilot study of dynamic contrast enhanced magnetic resonance imaging (DCE-MRI, aka perfusion MRI) and diffusion-weighted MRI (DWI-MRI), herein referred to in combination as advanced MRI (aMRI) in the investigation of early tumor response to standard multi-dose, fractionated external beam radiotherapy (EBRT) of the pelvis given in the neoadjuvant setting concurrent with chemotherapy as well as induction chemotherapy prior to chemoradiotherapy or consolidation chemotherapy after chemoradiotherapy for primary rectal adenocarcinoma. This protocol aims to expand upon the growing body of knowledge concerning early changes in tumor neovascularity and cellular density as a potential biomarker of therapy efficacy. It further aims to address the trend towards more refined treatment stratification for lower risk tumors to avoid morbidity from potentially unnecessary radiation, chemotherapy or even radical surgery, by assessing the earliest changes that occur in microvasculature and perfusion and diffusion of water during this treatment to see if these can be predictive of long-term efficacy of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary locally advanced rectal adenocarcinoma (0-18cm from the anal verge) confirmed by MSKCC pathologist and eligible to undergo chemoradiation and surgical resection at MSKCC.
* Written informed consent
* Age equal to or greater than 21 years
* Willing and able to undergo all study procedures
* Patients must have a planned surgical resection of the rectum

Exclusion Criteria:

* Patients younger than 21 years
* Pregnant and nursing women
* Contraindications for MRI (such as claustrophobia, pacemaker, non MR-compatible artificial heart valves, cochlear implants, surgical clips in the brain, metal fragments in eye)
* Estimated GFR (using Cockcroft formula Appendix 2) less than 30 ml/min/1.73m2 (FDA advises caution in using gadolinium-based contrast agents in patients with severe renal impairment).
* History of allergic reaction to MR contrast media
* Inability to give informed consent in person

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-04-09 (Actual); Primary Completion 2017-06-20 (Actual); Study Completion 2017-06-20 (Actual)

PRIMARY OUTCOMES:
determine the best MR imaging schedule | 3 years
  of early and midterm imaging times using DWI-MRI which will distinguish between near complete (90-99%)/complete pathology and clinical responders and partial/non-responders

SECONDARY OUTCOMES:
Determine if the best imaging schedule for DCE is the same as for DWI | 3 years
  The analysis plan will be identical to the one for the primary endpoint: six change measures will be computed for each DCE-MRI parameter (parameters Ktrans, Ve, kep, AUC 90, AUC 180) and each of these change measures will be evaluated as a predictor using the reference standard nCR/CR. ROC curves and the area under them will be estimated and used to rank the predictors.

CONTACTS AND LOCATIONS:
Overall Officials: Marc J. Gollub, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/